CLINICAL TRIAL: NCT01010230
Title: Vibration Intervention For Bone Enhancement In Childhood Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Gabrielle's Angel Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIBE; R21HD059292 (NIH); Gabrielle's Angel Fdn (Other: Gabrielle's Angel Foundation)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-04

CONDITIONS: Bone Mineral Density; Bone Strength
Keywords: Childhood cancer survivors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LMHF mechanical stimulation placebo device (Placebo Comparator): The placebo device is identical in appearance and function to the active platform; except when activated, it emits the same sound as the active device but does not deliver the vibration.
  Interventions: Device: LMHF mechanical stimulation placebo device
- LMHF mechanical stimulation (Active Comparator): Low magnitude, high frequency mechanical stimulation device ("vibrating") platform
  Interventions: Device: LMHF mechanical stimulation active device

INTERVENTIONS:
Device: LMHF mechanical stimulation active device — Participants will be randomly assigned to stand on a low magnitude, high frequency mechanical stimulation device ("vibrating") platform for 10 minutes twice daily for one year. The study hypothesizes participants in the intervention arm intervention will demonstrate improved total bone mineral content for height, spinal and tibial bone mineral density and tibial bone strength when compared to those who are randomized to the placebo intervention.
  Other Names: Bone mineral density
  Arms: LMHF mechanical stimulation
Device: LMHF mechanical stimulation placebo device — Participants will be randomly assigned to stand on a low magnitude, high frequency mechanical stimulation device ("vibrating") platform for 10 minutes twice daily for one year. The study hypothesizes participants in the intervention arm intervention will demonstrate improved total bone mineral content for height, spinal and tibial bone mineral density and tibial bone strength when compared to those who are randomized to the placebo intervention.
  Arms: LMHF mechanical stimulation placebo device

SUMMARY:
Treatment for childhood cancer interferes with normal bone maturation such that maximal peak bone mass may never be attained by some survivors of childhood cancer. In childhood cancer survivors, a randomized trial evaluating the effectiveness of vitamin D and calcium supplementation among ALL survivors is currently underway; however, few other interventions have been offered for this at risk population. Recent evidence demonstrates that low magnitude; high frequency mechanical stimulation can improve bone quantity and quality, perhaps providing an alternative or adjunct to pharmacologic intervention in populations where additional medications are either contraindicated or not acceptable to the individuals at risk. This application proposes a prospective double blind randomized clinical trial of low magnitude, high frequency mechanical (LMHF) stimulation for childhood cancer survivors whose bone mineral density is one or more standard deviations below the mean for their age and gender.

DETAILED DESCRIPTION:
This study is a two arm parallel allocation of participants to either the intervention or control group will be utilized for a one year trial.

Participants will be randomly assigned to stand on a low magnitude, high frequency mechanical stimulation device ("vibrating") platform for 10 minutes twice daily for one year. Participants in the control arm will stand on a placebo device.

This study will evaluate the effects of low magnitude, high frequency stimulus on bone mineral content(BMC), bone mineral density (BMD), and bone strength in childhood cancer survivors who present with BMD values 1.0 or more standard deviations below the mean for their age and gender for the lumbar or whole body. This study will evaluate the effects of low magnitude, high frequency stimulus on markers of bone turnover in childhood cancer survivors who present with BMD values 1.0 or more standard deviations below the mean for their age and gender for the lumbar or whole body.

At baseline participants will have evaluations to determine bone mineral content and bone mineral density (Dual X-ray Absorptiometry and Qualitative Computed Tomography) and a blood sample collected to measure biomarkers of bone turnover, hormonal status and Vitamin D metabolism. Anthropometrics and tanner stage will be obtained at baseline, 3 months, 6 months, 9 and 12 months. A physical activity monitor will be worn for a 7 day period and a food frequency questionnaire will be completed. Tibial length will be measured. Participants have a blood sample collected either at home or at St. Jude Children's Research Hospital (SJCRH) every 3 months during the study to measure biomarkers of bone turnover, hormonal status and Vitamin D metabolism, anthropometrics and tanner stage, physical activity monitor and food frequency questionnaire. All measurements and evaluations required at baseline will be repeated at the completion of study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Previously treated for childhood cancer at SJCRH
2. Greater than or equal to 5 years from childhood cancer diagnosis
3. Age and gender matched lumbar or whole body BMD z-score of <or equal -1.0
4. Not undergoing active treatment for cancer
5. ≥ 7 and <18 years of age
6. Able to stand for 10 minutes (May hold on to a support while standing)
7. Able to tolerate Calcium and Vitamin D supplements

Exclusion Criteria:

1. Receiving pharmacologic interventions other than Calcium and Vitamin D supplements for reduced Bone Mineral density (e.g. bisphosphonates)
2. Pregnant female
3. Individuals with metal implants that prevent BMD analysis by Dual X-ray Absorptiometry (DXA) or Quantitative Computed Tomography (QTC)
4. Inability or unwillingness of research participant or legal guardian/representative to give written informed consent/assent.
5. Spinal deformity requiring bracing
6. Chronic oral glucocorticoid therapy
7. Diagnosis of hereditary retinoblastoma (bilateral disease, familial, or positive test), Li-Fraumeni syndrome (positive testing for p53 mutation), Gorlin syndrome/Basil Cell Nevus syndrome, Bloom syndrome, Fanconi anemia, Ataxia telangiectasia or xeroderma pigmentosa

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2010-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten K Ness, PT, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Mogil RJ, Kaste SC, Ferry RJ Jr, Hudson MM, Mulrooney DA, Howell CR, Partin RE, Srivastava DK, Robison LL, Ness KK. Effect of Low-Magnitude, High-Frequency Mechanical Stimulation on BMD Among Young Childhood Cancer Survivors: A Randomized Clinical Trial. JAMA Oncol. 2016 Jul 1;2(7):908-14. doi: 10.1001/jamaoncol.2015.6557. PMID 26967465
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 81 participants enrolled 05/2010-10/2012. Each was: treated for childhood cancer, 5+ years from diagnosis, lumbar or whole body BMD z-scores of < -1.0, not currently being treated for cancer, 7-17 years, able to stand 10 min., tolerated calcium and vitamin-D supplements. Those with untreated endocrine disorders and pregnant females were excluded.
Pre-assignment Details: Fifteen participants were deemed ineligible after baseline testing, 11 because their bone density z-scores were > -1.0, one because they were on an oral steroid, one was older than the maximum age limit and two had unstable endocrine status. Two additional participants consented, but withdrew prior to baseline testing.
Groups:
- LMHF Mechanical Stimulation: Low magnitude, high frequency mechanical stimulation device ("vibrating") platform
  LMHF mechanical stimulation active device: Participants were randomly assigned to stand on a low magnitude, high frequency mechanical stimulation device ("vibrating") platform for 10 minutes twice daily for one year. The study hypothesized participants randomized to the active device would demonstrate improved total bone mineral content for height, spinal and tibial bone mineral density and tibial bone strength when compared to those who were randomized to the placebo intervention.
- Placebo Device: The placebo device is identical in appearance and function to the active platform; except when activated, it emits the same sound as the active device but does not deliver the vibration.
  Placebo device: Participants were randomly assigned to stand on a placebo device for 10 minutes twice daily for one year. The study hypothesized participants in the intervention arm would demonstrate improved total bone mineral content for height, spinal and tibial bone mineral density and tibial bone strength when compared to those who were randomized to the placebo arm.
Period: Overall Study
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Started | 32 | 33
Completed | 22 | 26
Not Completed | 10 | 7
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Population: The power estimates were based on two-sided two-sample t-tests. With 30 subjects in each of the two arms and assuming no change in the control arm (0% change) and assuming the common standard deviation (SD) of 6.8%3 we will have roughly 87% power to detect an improvement of 5.5% change in the intervention arm, with type I error control α=0.05.
Groups:
- Total: Total of all reporting groups
Arm/Group | LMHF Mechanical Stimulation | Placebo Device | Total
Number analyzed (Participants) | 22 | 26 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (2.7) | 13.5 (2.8) | 13.5 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Total Bone Mineral Content (BMC) Per Height Compared Between Intervention and Placebo Groups
Description: Since this is considered a "pilot study" we did not adjust for multiple comparisons. These % changes were treated as continuous variables and analyzed using two way ANOVAs adjusting for stratification.
Time Frame: Baseline and 12 months after start of intervention
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: % change in grams/cm
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
% change in grams/cm | 2.72 (10.41) | 3.96 (11.31)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; The power estimates were based on two-sided two-sample t-tests. With 30 subjects in each of the two arms and assuming no change in the control arm (0% change) and assuming the common standard deviation (SD) of 6.8% we estimated 87% power to detect an improvement of 5.5% change in the intervention arm, with type I error control α=0.05; Test type: Superiority or Other; p = 0.69, ANOVA — The threshold for significance was established a priori at alpha=0.05; BMC was normalized for height and adjusted for sex and tanner stage; Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-5.59 to 3.11]

2. Secondary Outcome: Mean Change in Aminoterminal Propeptide of Type I Procollagen (PINP) Compared Between the Intervention and Placebo Groups
Description: Biological markers of bone formation and cytokines collected at baseline and 12 months were evaluated to see if there was change over time.
Time Frame: Baseline and 12 months after the intervention begins
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: log of µg/L
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
log of µg/L | -0.11 (0.51) | -0.29 (0.34)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; Active and placebo group means were compared with a 2-sample t-test after log-transforming the variable; Test type: Non-Inferiority or Equivalence — The power calculation was based on the primary aim and is provided above; p = 0.18, t-test, 2 sided — The threshold for significance was established a priori at alpha=0.05; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [0.00 to 0.35]

3. Primary Outcome: Percent Change in Lumbar Spine Bone Mineral Content (BMC) Compared Between Intervention and Placebo Groups
Description: as for outcome 1
Time Frame: Baseline and 12 months after start of intervention/
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: % change in grams/cm
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
% change in grams/cm | 3.70 (21.15) | 2.54 (21.09)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.85, ANOVA — The threshold for significance was established a priori at alpha=0.05; BMC was normalized for height and adjusted for sex and tanner stage; Mean Difference (Final Values) = 1.16, 95% CI 2-sided [-6.93 to 9.25]

4. Primary Outcome: Percent Change in Total Bone Mineral Density (BMD) Compared Between Intervention and Placebo Groups
Description: as for outcome 1
Time Frame: Baseline and 12 months after the intervention begins
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: % change in g/cm^2
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
% change in g/cm^2 | 7.08 (10.20) | 4.88 (6.90)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; The power estimates were based on two-sided two-sample t-tests. With 30 subjects in each of the two arms and assuming no change in the control arm (0% change) and assuming the common standard deviation (SD) of 6.8%3 we estimated 87% power to detect an improvement of 5.5% change in the intervention arm, with type I error control α=0.05; Test type: Superiority or Other; p = 0.12, ANOVA — The threshold for significance was established a priori at alpha=0.05; Adjusted for sex and tanner stage; Mean Difference (Final Values) = 3.19, 95% CI 2-sided [0.43 to 5.95]

5. Primary Outcome: Percent Change in Lumbar Spine Bone Mineral Density (BMD) Compared Between Intervention and Placebo Groups
Description: as for outcome 1
Time Frame: Baseline and 12 months after the intervention begins
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: % change in g/cm^2
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
% change in g/cm^2 | 4.91 (10.34) | 5.01 (10.29)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.97, ANOVA — The threshold for significance was established a priori at alpha=0.05; Adjusted for sex and tanner stage (from general linear model); Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-4.24 to 4.05]

6. Primary Outcome: Percent Change in Lumbar Spine Volumetric Bone Mineral Density (BMD) Compared Between Intervention and Placebo Groups
Description: as for outcome 1
Time Frame: Baseline and 12 months after the intervention begins
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: % change in mg/cc
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
% change in mg/cc | 5.64 (10.83) | 5.30 (11.06)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.91, ANOVA — The threshold for significance was established a priori at alpha=0.05; Adjusted for sex and tanner stage; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-4.05 to 4.68]

7. Primary Outcome: Percent Change in Tibial Cortical Bone Compared Between the Intervention and Placebo Groups
Description: as for outcome 1
Time Frame: Baseline and 12 months after the intervention begins
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: % change in mg/cc
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
% change in mg/cc | 3.00 (4.69) | 1.77 (4.90)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.40, ANOVA — The threshold for significance was established a priori at alpha=0.05; Adjusted for sex and tanner stage; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [-0.69 to 3.11]

8. Primary Outcome: Percent Change in Cortical Bone Per Length Compared Between the Intervention and Placebo Groups
Description: as for outcome 1
Time Frame: Baseline and 12 months after the intervention begins
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: % change in mg/cm^4
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
% change in mg/cm^4 | -1.19 (6.63) | -1.86 (6.77)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.73, ANOVA — The threshold for significance was established a priori at alpha=0.05; Adjusted for sex and tanner stage; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [-2.02 to 3.33]

9. Secondary Outcome: Mean Change in Osteocalcin (OC) Compared Between the Intervention and Placebo Groups
Description: as for outcome 2
Time Frame: Baseline and 12 months after the intervention begins
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: log of ng/mL
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
log of ng/mL | -0.06 (0.30) | -0.27 (0.41)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; Active and placebo group means were compared with a 2-sample t-test after log-transforming the variable; Test type: Non-Inferiority or Equivalence — The power calculation was based on the primary aim and is provided above; p = 0.08, t-test, 2 sided — The threshold for significance was established a priori at alpha=0.05; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [0.06 to 0.34]

10. Secondary Outcome: Mean Change in Alkaline Phosphatase (ALP)-Skeletal (Bone Specific) Compared Between the Intervention and Placebo Groups
Description: as for outcome 2
Time Frame: Baseline and 12 months after the intervention begins
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: log of µg/L
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
log of µg/L | -0.18 (0.34) | -0.31 (0.30)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; Active and placebo group means were compared with a 2-sample t-test after log-transforming the variable; Test type: Non-Inferiority or Equivalence — The power calculation was based on the primary aim and is provided above; p = 0.17, t-test, 2 sided — The threshold for significance was established a priori at alpha=0.05; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [0.00 to 0.26]

11. Secondary Outcome: Mean Change in Carboxyterminal Telopeptide of Type I Collagen (ITCP) Compared Between the Intervention and Placebo Groups
Description: as for outcome 2
Time Frame: Baseline and 12 months after the intervention begins
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: log of µg/l
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
log of µg/l | -0.11 (0.30) | -0.19 (0.31)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; Active and placebo group means were compared with a 2-sample t-test after log-transforming the variable; Test type: Non-Inferiority or Equivalence — The power calculation was based on the primary aim and is provided above; p = 0.38, t-test, 2 sided — The threshold for significance was established a priori at alpha=0.05; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.04 to 0.20]

12. Secondary Outcome: Mean Change in Collagen Cross Linked N-Telepeptide (NTx) Compared Between the Intervention and Placebo Groups
Description: Biological markers of bone formation and cytokines collected at baseline and 12 months were evaluated to see if there was change over time. BCE = Bone Collagen Equivalent.
Time Frame: Baseline and 12 months after the intervention begins
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: log of 10 nmol BCE/L
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
log of 10 nmol BCE/L | -0.30 (0.56) | -0.28 (0.43)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; Active and placebo group means were compared with a 2-sample t-test after log-transforming the variable; Test type: Non-Inferiority or Equivalence — The power calculation was based on the primary aim and is provided above; p = 0.88, t-test, 2 sided — The threshold for significance was established a priori at alpha=0.05; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.22 to 0.18]

13. Secondary Outcome: Mean Change in Bone Turnover Ratio (RANKL/OPG) Compared Between the Intervention and Placebo Groups
Description: Biological markers evaluated are: Osteoprotegerin (OPG)/receptor activator nuclear factor kB ligand (sRANKL) index.
  Between-group comparisons used two-sample t-tests. Biomarkers and cytokines collected at baseline and 12 months were evaluated to see if there was change over time. Variables were log transformed for analysis.
Time Frame: Baseline and 12 months after the intervention begins
Population: This was an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: ratio of RANKL/OPG
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Number analyzed (Participants) | 22 | 26
ratio of RANKL/OPG | 0.14 (0.44) | -0.14 (0.50)
Statistical Analysis 1: Comparison: LMHF Mechanical Stimulation vs Placebo Device; Active and placebo group means were compared with a 2-sample t-test after log-transforming the variable; Test type: Non-Inferiority or Equivalence — The power calculation was based on the primary aim and is provided above; p = 0.06, t-test, 2 sided — The threshold for significance was established a priori at alpha=0.05; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [0.09 to 0.46]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the on-study date until 12 months after the start of intervention.
Description: Adverse events were reported in real time. The SJCRH IRB requires that study PI's report any unanticipated events involving risk to subjects or others during the conduct of the study. Appropriate action is discussed and the PI is notified to implement the decided action plan.
Arm/Group | LMHF Mechanical Stimulation | Placebo Device
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/26
Other Adverse Events (participants affected / at risk) | 0/22 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMHF Mechanical Stimulation (N=22) | Placebo Device (N=26)
Appendectomy (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Dropout was higher than expected leading to small numbers for analysis. It was estimated that 30 persons were needed in each arm to detect a 5.5% difference in change in bone outcomes between the active device and placebo device arms of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes